CLINICAL TRIAL: NCT04146987
Title: Cost-Effectiveness of Rotator Cuff Repair Surgery by Open and Arthroscopic Techniques. Randomized Clinical Trial
Brief Title: Cost-Effectiveness of Rotator Cuff Repair Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Hospital Alvorada (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 032019
Record Dates: First submitted 2019-10-14; First posted 2019-10-31 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-07

CONDITIONS: Rotator Cuff Injuries; Shoulder Pain; Shoulder Impingement; Shoulder Injuries; Shoulder Bursitis; Shoulder Tendinitis; Shoulder Lesions
Keywords: Rotator Cuff; Rotator Cuff Tear; Rotator Cuff Tendinopathy; Shoulder Arthroscopy; Rotator Cuff Repair; Open Rotator Cuff Repair
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain; Shoulder Impingement Syndrome; Shoulder Injuries

STUDY DESIGN:
Intervention Model Description: Patients will undergo a clinical evaluation, plain radiography, and magnetic resonance imaging to confirm the diagnosis of rotator cuff injury. At this moment, the type of lesion will be evaluated, as well as its size, retraction and the degree of fatty infiltration of the muscular belly, according to the Goutallier classification. The lesions will be classified as small (<1cm); moderate (1-3cm); large (3-5cm) or very large (> 5cm). All patients will undergo examinations and preoperative clinical evaluation.
  Patients will be consecutively allocated to one of two proposed treatment methods: open rotator cuff repair or arthroscopic rotator cuff repair.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Outcome evaluators will be masked (blinded) and not involved with the study. The statisticians who will conduct the analyzes will also be masked to the treatment status until the analyzes are completed. Due to the types of interventions, it will not be possible to mask the participants and providers of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open rotator cuff repair (Active Comparator): Patients will be positioned in a beach chair position with the affected limb pending off the table, allowing manipulation and full range of motion range. After asepsis, antisepsis and placement of sterile surgical fields, anterolateral incision will be made in the shoulder in question; the deltoid muscle belly will be gently divided along its fibers until exposure of the subdeltoid / subacromial bursa, which will be partially excised for exposure of the subacromial space and rotator cuff tendons. After mobilization and release of the ruptured tendons and debridement of the rotator cuff footprint, the tendon repair to the bone will be performed using 5.5m metal anchors, according to the preference and technique chosen by the surgeon. In all cases, the release of the coracoacromial ligament and acromioplasty will be performed.
  Interventions: Procedure: Rotator cuff repair surgery
- Arthroscopic rotator cuff repair (Active Comparator): The patients will be positioned in lateral decubitus position, with the arm to be operated attached to a skin traction device, which trough a traction post and 07 kg, will maintain the shoulder in the following position: abduction of 30 to 60 and flexion of 20 to 30 degrees. After asepsis, antisepsis and placement of impermeable sterile surgical fields, a posterolateral incision will be made in the shoulder for optic introduction, with a 50 mmHg pressure pump and a 0.90 flow, and inspection of the GU joint. After joint inspection, the optic will be introduced into the subacromial space with detachment of the subacromial and subdeltoid. Using shaver blades, partial bursectomy will be performed as well as debridement of the rotator cuff footprint. The tendon will then be reinserted to the bone using metallic 5.5mm anchors. After tendon repair, the coracoacromomial ligament will be released, as well as acromioplasty.
  Interventions: Procedure: Rotator cuff repair surgery

INTERVENTIONS:
Procedure: Rotator cuff repair surgery — Patients will undergo open rotator cuff repair or arthroscopic rotator cuff repair

SUMMARY:
Shoulder pain is one of the most common musculoskeletal complaints in orthopedic practice. Rotator cuff injuries account for up to 70% of pain in the shoulder girdle. There is no clinical study carried out in Brazil comparing cost effectiveness between the open and arthroscopic methods of rotator cuff repair surgery.

The present study aims to determine which method of repair of the rotator cuff, open or arthroscopic, has the best cost effectiveness ratio.

A randomized clinical trial will be carried out in which patients with symptomatic rotator cuff lesion will be submitted to repair surgery by either open or arthroscopic technique and will be subsequently evaluated.

DETAILED DESCRIPTION:
Introduction:

Musculoskeletal injuries are a major cost to the healthcare system. In 2004, 30% of the North American population had some kind of musculoskeletal disorder that required medical treatment; between 2002 and 2004, the estimated cost of treating these changes was $ 510 billion. Shoulder diseases represent the third most common cause of these changes, behind only spinal and knee disorders.

An evaluation of the primary health care system in Cambridge, United Kingdom, showed that the average frequency of shoulder pain was 9.5 per 1,000 individuals. Of these, 86% had rotator cuff tendinopathy. North American data estimate that approximately 4.5 million patients annually seek medical attention due to shoulder pain; of these, two million have some symptoms related to the rotator cuff. About 250,000 rotator cuff repair surgeries are performed annually in the United States of America (US), and with the continued increase in life expectancy and aging, there is a tendency to increase this number.

The rotator cuff is composed of the tendons of the subscapularis, supraspinatus, infraspinatus and teres minor muscles. The long portion of the biceps tendon also contributes to cuff function, which is to stabilize the humeral head in the glenoid cavity, preventing superior migration of the humeral head.

The possible lesions range from tendon degeneration (tendinosis/tendinopathy), through partial lesions (articular, interstitial or bursal), to complete lesions. Diagnosis is made by associating history and physical examination along with imaging methods, and magnetic resonance imaging (MRI) is considered the method of choice.

Currently, the indication for surgical treatment is based on the persistence of symptoms and/or the degree of muscle weakness and/or size of the lesion, after a time of conservative treatment. In general, when opting for surgery, imaging can assist in the planning of surgical treatment, since it allows measuring the extent of the lesion (partial or total) and discriminating which tendons are involved (supraspinatus, infraspinatus, etc.).

Treatment of rotator cuff diseases depends on the type of injury, the patient's degree of activity, age, and the presence of symptoms. In general, tendon degeneration and partial lesions are treated non-surgically, with physiotherapy, infiltrations and analgesic medications. Complete and incomplete lesions that did not respond well to conservative treatment, however, should be treated surgically. Among the surgical options, the open method is still considered the gold standard, with good or excellent results in over 90% of cases. With the advent of arthroscopy and the evolution of arthroscopic instruments and implants in the last decade, the arthroscopic repair technique has gained space and is widely used in the investigator's country. Several studies abroad did not demonstrate superiority of one technique over another in terms of clinical outcomes. As the cost of arthroscopic surgery is higher, due to the equipment needed to perform it, it is important to establish which option has the best cost-effectiveness.

Some studies abroad even suggest the superiority of the open method over the arthroscopic method. However, there are no studies comparing cost-effectiveness between open and arthroscopic methods in Brazil. Therefore, the present study aims to compare the open and arthroscopic methods for rotator cuff repair and determine which presents the best cost-effectiveness ratio.

Hypothesis:

The hypothesis of this study is that the open method of rotator cuff repair will be more cost-effective compared to the arthroscopic method.

Justification:

In a systematic literature search, it was observed that there are no studies in the Brazilian literature comparing the cost-effectiveness of open and arthroscopic rotator cuff repair methods. Data from the international literature suggest that the open repair method is more cost-effective than the arthroscopic method (same clinical outcome and lower cost).

Thus, despite the high incidence of rotator cuff injury, there is insufficient evidence from the Brazilian experience to determine the best method for treating these injuries. So, this project proposes to conduct a study to answer the clinical question of which method, open or arthroscopic, has the best cost-effectiveness in the surgical treatment of rotator cuff injury. According to the levels of scientific evidence, the most appropriate study design to answer this clinical question is a randomized clinical trial.

Study Goal:

The present study aims to compare the open and arthroscopic methods for rotator cuff repair and determine which presents the best cost-effectiveness ratio.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complete rotator cuff injury, symptomatic, where there was failure or the patient could not support the non-surgical treatment;
* Patients with high-grade partial rotator cuff injury where therapy failed or the patient did not support non-surgical treatment;
* Patients without medical contraindications for surgery;
* Patients with a good understanding of the Portuguese language and who agree to participate and sign the Informed Consent Form.

Exclusion Criteria:

* Patients under 18 years old
* Patients with previous shoulder surgery;
* Patients with limited range of motion of the shoulder (joint stiffness);
* Patients with previous fractures in the affected shoulder;
* Patients with signs of glenohumeral osteoarthritis;
* Patients with neurological injury;
* Patients who opt not to participate and/or are not willing to sign the informed consent form;
* Patients unable to complete the follow-up evaluation (inability to read or complete the forms).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Constant-Murley Score (CM) | Measured continuously for 48 weeks after the intervention
  The Constant-Murley Score (CM) validated for the Portuguese language. The evaluators will ask the patients to fill in the validated CM form for the Portuguese language and measure the range of motion with a goniometer. The CM scale covers different domains of shoulder function (pain, activities of daily living, range of motion and power), punctuating each of them; it ranges from 0 to 100, with higher scores indicating better function.
EuroQol-5D-3L (European Quality of Life) | Measured continuously for 48 weeks after the intervention
  EuroQol-5D-3L (European Quality of Life), a generic score developed to describe health-related quality of life will also be assessed preoperatively, at 6, 24 and 48 weeks postoperatively. This score includes five health domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression; each domain has 3 levels: no problem; some problems and extreme problems. In addition, the EuroQol-5D-3L has a visual analog scale where the participant assigns a value between zero and one hundred to his or her own health condition. At the end of its application, EuroQol-5D-3L will provide a unique numerical value that can be used for longitudinal comparison between two time periods (pre and postoperative, for example).

SECONDARY OUTCOMES:
Simple Shoulder Test (SST) | Measured continuously for 48 weeks after the intervention
  SST is a simple, quick and widely used questionnaire for shoulder function measurement; it consists of 12 dichotomous questions answered by the patient himself. Each positive answer (yes) is given a score; at the end of the questionnaire the percentage of positive answers (score) is made, and the higher the percentage, the better the shoulder function.
Visual Analogue Pain Scale (VAS) | Measured continuously for 48 weeks after the intervention
  This scale allows pain intensity to be measured with maximum interobserver reproducibility; it consists of a 10 cm straight line with the ends determining the limits of pain sensation (no pain; worst pain ever experienced); the distance between zero (no pain) and the patient's demarcation defines the intensity of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Pierami, MD, Principal Investigator — SOCIEDADE BENEF ISRAELITABRAS HOSPITAL ALBERT EINSTEIN
Locations (2):
- Brazil (2):
  - Hospital Alvorada Moema, São Paulo, São Paulo
  - Hospital Israelita Albert Einstein (HIAE), São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mather RC 3rd, Koenig L, Acevedo D, Dall TM, Gallo P, Romeo A, Tongue J, Williams G Jr. The societal and economic value of rotator cuff repair. J Bone Joint Surg Am. 2013 Nov 20;95(22):1993-2000. doi: 10.2106/JBJS.L.01495. PMID 24257656
- [Result] Kuye IO, Jain NB, Warner L, Herndon JH, Warner JJ. Economic evaluations in shoulder pathologies: a systematic review of the literature. J Shoulder Elbow Surg. 2012 Mar;21(3):367-75. doi: 10.1016/j.jse.2011.05.019. Epub 2011 Aug 23. PMID 21865060
- [Result] Ostor AJ, Richards CA, Prevost AT, Speed CA, Hazleman BL. Diagnosis and relation to general health of shoulder disorders presenting to primary care. Rheumatology (Oxford). 2005 Jun;44(6):800-5. doi: 10.1093/rheumatology/keh598. Epub 2005 Mar 15. PMID 15769790
- [Result] Favard L, Bacle G, Berhouet J. Rotator cuff repair. Joint Bone Spine. 2007 Dec;74(6):551-7. doi: 10.1016/j.jbspin.2007.08.003. Epub 2007 Oct 12. PMID 17993287
- [Result] Tempelaere C, Pierrart J, Lefevre-Colau MM, Vuillemin V, Cuenod CA, Hansen U, Mir O, Skalli W, Gregory T. Dynamic Three-Dimensional Shoulder Mri during Active Motion for Investigation of Rotator Cuff Diseases. PLoS One. 2016 Jul 19;11(7):e0158563. doi: 10.1371/journal.pone.0158563. eCollection 2016. PMID 27434235
- [Result] Sela Y, Eshed I, Shapira S, Oran A, Vogel G, Herman A, Perry Pritsch M. Rotator cuff tears: correlation between geometric tear patterns on MRI and arthroscopy and pre- and postoperative clinical findings. Acta Radiol. 2015 Feb;56(2):182-9. doi: 10.1177/0284185114520861. Epub 2014 Jan 20. PMID 24445094
- [Result] Teefey SA, Rubin DA, Middleton WD, Hildebolt CF, Leibold RA, Yamaguchi K. Detection and quantification of rotator cuff tears. Comparison of ultrasonographic, magnetic resonance imaging, and arthroscopic findings in seventy-one consecutive cases. J Bone Joint Surg Am. 2004 Apr;86(4):708-16. PMID 15069134
- [Result] Jason E. Hsu Steven B. Lippitt, Frederick A. Matsen III AOG. Rockwood and Matsen's The Shoulder, 5th Edition: The Rotator Cuff. In: Rockwood and Matsen's The Shoulder, 5th Edition. 5th ed. Elsevier; 2016. p. 651-719.
- [Result] Yamakawa S, Hashizume H, Ichikawa N, Itadera E, Inoue H. Comparative studies of MRI and operative findings in rotator cuff tear. Acta Med Okayama. 2001 Oct;55(5):261-8. doi: 10.18926/AMO/32019. PMID 11688948
- [Result] Roy JS, Braen C, Leblond J, Desmeules F, Dionne CE, MacDermid JC, Bureau NJ, Fremont P. Diagnostic accuracy of ultrasonography, MRI and MR arthrography in the characterisation of rotator cuff disorders: a systematic review and meta-analysis. Br J Sports Med. 2015 Oct;49(20):1316-28. doi: 10.1136/bjsports-2014-094148. Epub 2015 Feb 11. PMID 25677796
- [Result] Lenza M, Buchbinder R, Takwoingi Y, Johnston RV, Hanchard NC, Faloppa F. Magnetic resonance imaging, magnetic resonance arthrography and ultrasonography for assessing rotator cuff tears in people with shoulder pain for whom surgery is being considered. Cochrane Database Syst Rev. 2013 Sep 24;2013(9):CD009020. doi: 10.1002/14651858.CD009020.pub2. PMID 24065456
- [Result] Handoll HH, Hanchard NC, Lenza M, Buchbinder R. Rotator cuff tears and shoulder impingement: a tale of two diagnostic test accuracy reviews. Cochrane Database Syst Rev. 2013 Oct 7;2013(10):ED000068. doi: 10.1002/14651858.ED000068. No abstract available. PMID 24475489
- [Result] Hanchard NC, Lenza M, Handoll HH, Takwoingi Y. Physical tests for shoulder impingements and local lesions of bursa, tendon or labrum that may accompany impingement. Cochrane Database Syst Rev. 2013 Apr 30;2013(4):CD007427. doi: 10.1002/14651858.CD007427.pub2. PMID 23633343
- [Result] Seida JC, LeBlanc C, Schouten JR, Mousavi SS, Hartling L, Vandermeer B, Tjosvold L, Sheps DM. Systematic review: nonoperative and operative treatments for rotator cuff tears. Ann Intern Med. 2010 Aug 17;153(4):246-55. doi: 10.7326/0003-4819-153-4-201008170-00263. Epub 2010 Jul 5. PMID 20621893
- [Result] Ainsworth R, Lewis JS. Exercise therapy for the conservative management of full thickness tears of the rotator cuff: a systematic review. Br J Sports Med. 2007 Apr;41(4):200-10. doi: 10.1136/bjsm.2006.032524. Epub 2007 Jan 30. PMID 17264144
- [Result] Eljabu W, Klinger HM, von Knoch M. The natural history of rotator cuff tears: a systematic review. Arch Orthop Trauma Surg. 2015 Aug;135(8):1055-61. doi: 10.1007/s00402-015-2239-1. Epub 2015 May 6. PMID 25944157
- [Result] van der Zwaal P, Thomassen BJ, Nieuwenhuijse MJ, Lindenburg R, Swen JW, van Arkel ER. Clinical outcome in all-arthroscopic versus mini-open rotator cuff repair in small to medium-sized tears: a randomized controlled trial in 100 patients with 1-year follow-up. Arthroscopy. 2013 Feb;29(2):266-73. doi: 10.1016/j.arthro.2012.08.022. Epub 2012 Dec 1. PMID 23206691
- [Result] Morse K, Davis AD, Afra R, Kaye EK, Schepsis A, Voloshin I. Arthroscopic versus mini-open rotator cuff repair: a comprehensive review and meta-analysis. Am J Sports Med. 2008 Sep;36(9):1824-8. doi: 10.1177/0363546508322903. PMID 18753683
- [Result] Ji X, Bi C, Wang F, Wang Q. Arthroscopic versus mini-open rotator cuff repair: an up-to-date meta-analysis of randomized controlled trials. Arthroscopy. 2015 Jan;31(1):118-24. doi: 10.1016/j.arthro.2014.08.017. Epub 2014 Oct 16. PMID 25442664
- [Result] Huang R, Wang S, Wang Y, Qin X, Sun Y. Systematic Review of All-Arthroscopic Versus Mini-Open Repair of Rotator Cuff Tears: A Meta-Analysis. Sci Rep. 2016 Mar 7;6:22857. doi: 10.1038/srep22857. PMID 26947557
- [Result] Adla DN, Rowsell M, Pandey R. Cost-effectiveness of open versus arthroscopic rotator cuff repair. J Shoulder Elbow Surg. 2010 Mar;19(2):258-61. doi: 10.1016/j.jse.2009.05.004. Epub 2009 Jul 1. PMID 19574063
- [Result] Kose KC, Tezen E, Cebesoy O, Karadeniz E, Guner D, Adiyaman S, Demirtas M. Mini-open versus all-arthroscopic rotator cuff repair: comparison of the operative costs and the clinical outcomes. Adv Ther. 2008 Mar;25(3):249-59. doi: 10.1007/s12325-008-0031-0. PMID 18363045
- [Result] Vitale MA, Vitale MG, Zivin JG, Braman JP, Bigliani LU, Flatow EL. Rotator cuff repair: an analysis of utility scores and cost-effectiveness. J Shoulder Elbow Surg. 2007 Mar-Apr;16(2):181-7. doi: 10.1016/j.jse.2006.06.013. PMID 17399623
- [Result] Hui YJ, Teo AQ, Sharma S, Tan BH, Kumar VP. Immediate costs of mini-open versus arthroscopic rotator cuff repair in an Asian population. J Orthop Surg (Hong Kong). 2017 Jan;25(1):2309499016684496. doi: 10.1177/2309499016684496. PMID 28193144
- [Result] Churchill RS, Ghorai JK. Total cost and operating room time comparison of rotator cuff repair techniques at low, intermediate, and high volume centers: mini-open versus all-arthroscopic. J Shoulder Elbow Surg. 2010 Jul;19(5):716-21. doi: 10.1016/j.jse.2009.10.011. Epub 2010 Feb 4. PMID 20137974
- [Result] Altman DG, Schulz KF, Moher D, Egger M, Davidoff F, Elbourne D, Gotzsche PC, Lang T; CONSORT GROUP (Consolidated Standards of Reporting Trials). The revised CONSORT statement for reporting randomized trials: explanation and elaboration. Ann Intern Med. 2001 Apr 17;134(8):663-94. doi: 10.7326/0003-4819-134-8-200104170-00012. PMID 11304107
- [Result] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Result] Bhandari M, Guyatt GH, Swiontkowski MF. User's guide to the orthopaedic literature: how to use an article about prognosis. J Bone Joint Surg Am. 2001 Oct;83(10):1555-64. doi: 10.2106/00004623-200110000-00017. No abstract available. PMID 11679610
- [Result] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. Trials. 2010 Mar 24;11:32. doi: 10.1186/1745-6215-11-32. PMID 20334632
- [Result] DeOrio JK, Cofield RH. Results of a second attempt at surgical repair of a failed initial rotator-cuff repair. J Bone Joint Surg Am. 1984 Apr;66(4):563-7. PMID 6707035
- [Result] Goutallier D, Postel JM, Bernageau J, Lavau L, Voisin MC. Fatty muscle degeneration in cuff ruptures. Pre- and postoperative evaluation by CT scan. Clin Orthop Relat Res. 1994 Jul;(304):78-83. PMID 8020238
- [Result] Fuchs B, Weishaupt D, Zanetti M, Hodler J, Gerber C. Fatty degeneration of the muscles of the rotator cuff: assessment by computed tomography versus magnetic resonance imaging. J Shoulder Elbow Surg. 1999 Nov-Dec;8(6):599-605. doi: 10.1016/s1058-2746(99)90097-6. PMID 10633896
- [Result] Barreto RP, Barbosa ML, Balbinotti MA, Mothes FC, da Rosa LH, Silva MF. The Brazilian version of the Constant-Murley Score (CMS-BR): convergent and construct validity, internal consistency, and unidimensionality. Rev Bras Ortop. 2016 Oct 26;51(5):515-520. doi: 10.1016/j.rboe.2016.08.017. eCollection 2016 Sep-Oct. PMID 27818971
- [Result] Sanders GD, Neumann PJ, Basu A, Brock DW, Feeny D, Krahn M, Kuntz KM, Meltzer DO, Owens DK, Prosser LA, Salomon JA, Sculpher MJ, Trikalinos TA, Russell LB, Siegel JE, Ganiats TG. Recommendations for Conduct, Methodological Practices, and Reporting of Cost-effectiveness Analyses: Second Panel on Cost-Effectiveness in Health and Medicine. JAMA. 2016 Sep 13;316(10):1093-103. doi: 10.1001/jama.2016.12195. PMID 27623463
- [Result] Noronha F. Associação Portuguesa de Economia da Saúde Lara de Noronha e Ferreira. 2002;46
- [Result] Neto JO, Gesser RL, Steglich V, Bonilauri Ferreira AP, Gandhi M, Vissoci JR, Pietrobon R. Validation of the Simple Shoulder Test in a Portuguese-Brazilian population. Is the latent variable structure and validation of the Simple Shoulder Test Stable across cultures? PLoS One. 2013 May 13;8(5):e62890. doi: 10.1371/journal.pone.0062890. Print 2013. PMID 23675436
- [Result] D. G. Altman. Practical statistics for medical research. In: CRC Press. London; 1991
- [Result] Faraway JJ. Extending the linear model with R: generalized linear, mixed effects and nonparametric regression models. Taylor & Francis. 2006
- [Result] IBM Corp. Released 2016. IBM SPSS Statistics for Macintosh, Version 24.0. Armonk NIC. IBM Corp. Knowledge Management. 2005
- [Result] Kukkonen J, Kauko T, Vahlberg T, Joukainen A, Aarimaa V. Investigating minimal clinically important difference for Constant score in patients undergoing rotator cuff surgery. J Shoulder Elbow Surg. 2013 Dec;22(12):1650-5. doi: 10.1016/j.jse.2013.05.002. Epub 2013 Jul 12. PMID 23850308
- [Result] NCSS L. PASS 14 Power Analysis and Sample Size Software. Kaysville, Utah, USA; 2015.
- [Result] Sackett DL, Rosenberg WM, Gray JA, Haynes RB, Richardson WS. Evidence based medicine: what it is and what it isn't. BMJ. 1996 Jan 13;312(7023):71-2. doi: 10.1136/bmj.312.7023.71. No abstract available. PMID 8555924
- [Derived] Pierami R, Antonioli E, Oliveira I, Castro IQ, Manente F, Fairbanks P, Carrera EDF, Matsumura BA, Lenza M. Clinical outcomes and cost-utility of rotator cuff repair surgery by open and arthroscopic techniques: study protocol for a randomised clinical trial. BMJ Open. 2020 Dec 28;10(12):e043126. doi: 10.1136/bmjopen-2020-043126. PMID 33372080

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT04146987/Prot_SAP_000.pdf